CLINICAL TRIAL: NCT00784875
Title: A Phase 2, Randomized, Double-Blind, Placebo- and Active-Comparator-Controlled Study of the Safety and Efficacy of LY2624803 in Outpatients With Insomnia
Brief Title: An Efficacy Study of Compound LY2624803 in the Treatment of Patients With Chronic Insomnia
Acronym: SLUMBER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 12063; I2K-MC-ZZAD (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-10-31; First posted 2008-11-04 (Estimated); Results first posted 2012-02-29 (Estimated); Last update posted 2012-02-29 (Estimated); Status verified 2012-01

CONDITIONS: Primary Insomnia; Secondary Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Zolpidem

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Period A (Experimental): 2-week double-blind placebo lead-in period. Period A is the first of four 2-week treatment periods.
  Interventions: Drug: Placebo
- Period B (Experimental): Patients will receive LY2624803, zolpidem or placebo in a sequence of four 2-week treatment periods. Period B is the second of four 2-week treatment periods.
  Interventions: Drug: LY2624803; Drug: Placebo; Drug: zolpidem
- Period C (Experimental): Patients will receive LY2624803, zolpidem or placebo in a sequence of four 2-week treatment periods. Period C is the third of four 2-week treatment periods.
  Interventions: Drug: LY2624803; Drug: Placebo; Drug: zolpidem
- Period D (Experimental): Patients will receive LY2624803, zolpidem or placebo in a sequence of four 2-week treatment periods. Period D is the fourth of four 2-week treatment periods.
  Interventions: Drug: LY2624803; Drug: Placebo; Drug: zolpidem

INTERVENTIONS:
Drug: LY2624803 — 1 mg, oral capsule, once nightly before bedtime
  Arms: Period B; Period C; Period D
Drug: LY2624803 — 3 mg, oral capsule, once nightly before bedtime
  Arms: Period B; Period C; Period D
Drug: Placebo — matching placebo (capsule or tablet), once nightly before bedtime
Drug: zolpidem — 5 or 10 mg, oral tablet, once nightly before bedtime
  Arms: Period B; Period C; Period D

SUMMARY:
The purpose of this study is to compare an investigational drug (LY2624803) with placebo and with zolpidem in the treatment of outpatients with chronic insomnia.

DETAILED DESCRIPTION:
Outpatients with chronic insomnia who participate in this study will be treated in each of four 2-week treatment periods with bedtime doses of either placebo, zolpidem, LY2624803 1 mg, or LY2624803 3 mg. Neither patients nor investigators will be told what treatments are being given in any treatment period. A patient who completes all four treatment periods will be treated with placebo in 1, 2, or 3 of the periods; with zolpidem in 0, 1, or 2 of the periods; and with LY2624803 in either 1 or 2 of the periods. No patient will receive placebo for all four of the 2-week treatment periods. All patients will receive LY2624803 for at least one of the four 2-week treatment periods. During each treatment period, patients will record information each morning about their sleep the night before, and each evening about their functioning since waking up. Patients will also wear wrist actigraphy devices to record their physical activity. At the conclusion of each treatment period, patients will answer questions about their sleep, functioning, health, and relative preference for treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be between 18 and 85 years of age, with a stable living situation
* Clinical diagnosis of either primary insomnia or "secondary" insomnia (comorbid with depression, anxiety, and/or medical illness)
* Insomnia systems must be at least moderate in severity within the month prior to study entry, and must include difficulty staying asleep and/or problems with awakening earlier than desired
* Psychiatric and medical conditions present must be stable over the 3 months prior to study entry, and not expected to worsen significantly or require hospitalization during participation in the study
* Ongoing treatments for psychiatric and medical conditions present must have been stable for the 3 months prior to study entry, and must be expected to remain stable during participation in the study
* Patients must be willing to abstain from taking medications (other than study drug) to help them sleep during participation in the study
* Patients must be willing to consistently spend at least 7 hours each night either sleeping or trying to sleep during participation in the study
* Patients must be able to speak and read English and be capable of using a computer with a web browser (computers with internet connections will be provided to patients who need them)

Exclusion Criteria:

* Unusual or unstable sleep/wake schedule, such as with rotating shift work
* Severe or unstable psychiatric or medical illness
* Suicidal ideation
* Substance abuse
* Known obstructive sleep apnea, restless leg syndrome, or periodic limb movement disorder
* History of seizures
* Body Mass Index > 33
* Clinically significant abnormality in clinical chemistry, hematology, urinalysis, and/or electrocardiogram
* Anticipated inability to regularly use a medication which might reduce motor or cognitive functioning during sleeping hours, such as a person who might often need to be "on call", drive a car, or be responsible for the care of another person during sleeping hours
* Contraindication to zolpidem
* History of breast cancer
* An estimated glomerular filtration rate (GFR; an index of renal function) that is <30 mL/min at study entry

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 643 (Actual)
Dates: Start 2008-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (49):
- United States (49):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glendale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mesa, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Little Rock, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burbank, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glendale, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oceanside, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pismo Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Rosa, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torrance, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fruitland Park, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hialeah, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lauderdale Lakes, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Maitland, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Naples, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pembroke Pines, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St. Petersburg, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suwanee, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oak Brook, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Terre Haute, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Crestview Hills, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chevy Chase, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wellesley Hills, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sterling Heights, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Florissant, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brooklyn, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Bronx, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hickory, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Raleigh, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winston-Salem, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jenkintown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lincoln, Rhode Island
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Anderson, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bellevue, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lakewood, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: LY2624803 was placed on clinical hold by Food and Drug Administration (FDA) on 18 December 2008. The FDA lifted the clinical hold effective 05 May 2009. For analysis purposes, participants who entered into study during 2008 were designated as Cohort 1, whereas participants who entered into study after 2008 were designated as Cohort 2.
Pre-assignment Details: None of Cohort 1 participants completed the study and few progressed beyond Period B. The efficacy analyses were conducted using data from Cohort 2 participants only. Participant flow includes participants from both cohorts.
Groups:
- LY2624803 1 mg: Participants received LY2624803 1 mg in a 2-week treatment period.
- LY2624803 3 mg: Participants received LY2624803 3 mg in a 2-week treatment period.
- Zolpidem 5 or 10 mg: Participants received Zolpidem 5 or 10 mg in a 2-week treatment period.
- Placebo: Participants received placebo in a 2-week treatment period.
Period: Period A - Baseline
Arm/Group | LY2624803 1 mg | LY2624803 3 mg | Zolpidem 5 or 10 mg | Placebo
Started | 0 | 0 | 0 | 643
Completed | 0 | 0 | 0 | 461
Not Completed | 0 | 0 | 0 | 182
Not completed — Entry Criteria Not Met | 0 | 0 | 0 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 8
Not completed — Protocol Violation | 0 | 0 | 0 | 25
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 27
Not completed — Physician Decision | 0 | 0 | 0 | 2
Not completed — Sponsor Decision | 0 | 0 | 0 | 113
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2
Period: Period B - Efficacy Endpoint
Arm/Group | LY2624803 1 mg | LY2624803 3 mg | Zolpidem 5 or 10 mg | Placebo
Started | 114 | 113 | 117 | 117
Cohort 2 | 102 | 102 | 102 | 101
Completed | 100 | 101 | 96 | 98
Not Completed | 14 | 12 | 21 | 19
Not completed — Entry Criteria Not Met | 0 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 3 | 2 | 1
Not completed — Protocol Violation | 1 | 1 | 2 | 3
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 1 | 1 | 2
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Sponsor Decision | 9 | 6 | 12 | 12
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Period: Period C
Arm/Group | LY2624803 1 mg | LY2624803 3 mg | Zolpidem 5 or 10 mg | Placebo
Started | 103 | 97 | 97 | 98
Completed | 96 | 91 | 84 | 91
Not Completed | 7 | 6 | 13 | 7
Not completed — Adverse Event | 1 | 0 | 4 | 2
Not completed — Protocol Violation | 0 | 0 | 1 | 2
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 1
Not completed — Sponsor Decision | 5 | 5 | 4 | 2
Period: Period D
Arm/Group | LY2624803 1 mg | LY2624803 3 mg | Zolpidem 5 or 10 mg | Placebo
Started | 91 | 89 | 94 | 88
Completed | 86 | 85 | 88 | 87
Not Completed | 5 | 4 | 6 | 1
Not completed — Adverse Event | 0 | 2 | 2 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 2 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Sponsor Decision | 1 | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- LY2624803 1 mg: Participants received LY2624803 1 mg in Period B (2-week treatment period).
- LY2624803 3 mg: Participants received LY2624803 3 mg in Period B (2-week treatment period).
- Zolpidem 5 or 10 mg: Participants received Zolpidem 5 or 10 mg in Period B (2-week treatment period).
- Placebo: Participants received placebo in Period B (2-week treatment period).
- Total: Total of all reporting groups
Arm/Group | LY2624803 1 mg | LY2624803 3 mg | Zolpidem 5 or 10 mg | Placebo | Total
Number analyzed (Participants) | 102 | 102 | 102 | 101 | 407
Age Continuous [Mean (Standard Deviation); unit: years] | 52.81 (14.07) | 52.77 (14.73) | 50.65 (15) | 52.86 (13.66) | 52.27 (14.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 52 | 61 | 61 | 240
  Male | 36 | 50 | 41 | 40 | 167
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 75 | 74 | 85 | 72 | 306
  African | 21 | 21 | 12 | 18 | 72
  Hispanic | 6 | 5 | 3 | 9 | 23
  East Asian | 0 | 2 | 1 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 102 | 102 | 102 | 101 | 407

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Nightly Total Sleep Time at Week 4 (Week 2 of Period B) Endpoint
Description: Total Sleep Time is defined as time in bed minus total time awake. Minimum would be 0; no defined maximum (except if as defined as time in bed). The higher the number, the more time asleep. Calculated in minutes from participant-reported daily sleep questionnaire averaged across study Period B (2 weeks). Change score subtracts Period B average from Period A average (baseline). Analysis of covariance (ANCOVA) Model with dependent variable being change from baseline scores and independent variables being treatment, baseline, age group (<65 or ≥65), and insomnia type (primary vs. secondary).
Time Frame: Baseline, 2 weeks
Population: All randomized Cohort 2 participants who received at least one dose of study drug, and had both baseline and endpoint values.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | LY2624803 1 mg | LY2624803 3 mg | Zolpidem 5 or 10 mg | Placebo
Number analyzed (Participants) | 102 | 102 | 102 | 101
minutes | 30.16 (5.300) | 37.33 (5.186) | 50.63 (5.186) | 22.79 (5.153)

2. Secondary Outcome: Change From Baseline in Unwanted Time Awake at Week 4 (Week 2 of Period B) Endpoint
Description: Unwanted time awake (minutes awake [MA] before sleep [between turning off the lights to first falling asleep], MA during sleep, MA after sleep before getting out of bed). Minimum would be 0; no defined maximum. The higher the number, the more the unwanted time awake. Calculated in minutes from participant-reported daily sleep questionnaire averaged (Avg.) across Period B. Change score subtracts Period B Avg. from Period A Avg. (baseline). ANCOVA Model with dependent variable being change from baseline scores and independent variables being treatment, baseline, age group, and insomnia type.
Time Frame: Baseline, 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | LY2624803 1 mg | LY2624803 3 mg | Zolpidem 5 or 10 mg | Placebo
Number analyzed (Participants) | 102 | 102 | 102 | 101
minutes
  Before Sleep (n= 101, 101, 101, 101) | -7.08 (2.524) | -6.45 (2.444) | -20.48 (2.440) | -1.46 (2.420)
  During Sleep (n= 101, 102, 101, 101) | -14.84 (2.881) | -12.95 (2.812) | -21.46 (2.819) | -8.23 (2.794)
  After Sleep (n= 100, 101, 99, 99) | -9.07 (2.150) | -8.31 (2.108) | -4.91 (2.119) | -5.05 (2.105)

3. Secondary Outcome: Change From Baseline in Number of Awakenings During Sleep at Week 4 (Week 2 of Period B) Endpoint
Description: Elicited from participant-reported daily sleep questionnaire averaged across study Period B (2 weeks). Change score subtracts Period B average from Period A average (baseline). ANCOVA Model with dependent variable being change from baseline scores and independent variables being treatment, baseline, age group (<65 or ≥65), and insomnia type (primary vs. secondary).
Time Frame: Baseline, 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: number of awakenings
Arm/Group | LY2624803 1 mg | LY2624803 3 mg | Zolpidem 5 or 10 mg | Placebo
Number analyzed (Participants) | 102 | 102 | 102 | 101
number of awakenings | -0.27 (0.066) | -0.26 (0.065) | -0.59 (0.065) | -0.18 (0.065)

4. Secondary Outcome: Change From Baseline in Total Time Awake at Week 4 (Week 2 of Period B) Endpoint
Description: Calculated in minutes from participant-reported daily sleep questionnaire averaged across study Period B (2 weeks). Change score subtracts Period B average from Period A average (baseline). ANCOVA Model with dependent variable being change from baseline scores and independent variables being treatment, baseline, age group (<65 or ≥65), and insomnia type (primary vs. secondary).
Time Frame: Baseline, 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | LY2624803 1 mg | LY2624803 3 mg | Zolpidem 5 or 10 mg | Placebo
Number analyzed (Participants) | 102 | 102 | 102 | 101
minutes | -28.63 (4.678) | -28.62 (4.591) | -47.28 (4.579) | -13.09 (4.547)

5. Secondary Outcome: Change From Baseline in Sleep Efficiency at Week 4 (Week 2 of Period B) Endpoint
Description: Calculated as (TIB-TTA)/TIB where TIB is time in bed and TTA is total unwanted time awake. Higher score indicates better sleep efficiency. ANCOVA Model with dependent variable being change from baseline scores and independent variables being treatment, baseline, age group (<65 or ≥65), and insomnia type (primary vs. secondary).
Time Frame: Baseline, 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | LY2624803 1 mg | LY2624803 3 mg | Zolpidem 5 or 10 mg | Placebo
Number analyzed (Participants) | 102 | 102 | 102 | 101
ratio | 0.06 (0.009) | 0.06 (0.009) | 0.10 (0.009) | 0.03 (0.009)

6. Secondary Outcome: Change From Baseline in Assessment of Sleep Quality at Week 4 (Week 2 of Period B) Endpoint
Description: Assessment of Sleep Quality (ASQ) scale is asked in the participant-reported daily sleep questionnaire; 8 items on 4 point Likert scale with a range of 0 to 24. Sleep experience score ranges from 0-9; awakening experience ranges from 0-15. The higher the score, the better the sleep. Scale is averaged across study Period B (2 weeks). Change score subtracts Period B average from Period A average (baseline). ANCOVA Model with dependent variable being change from baseline scores and independent variables being treatment, baseline, age group (<65 or ≥65), and insomnia type (primary vs. secondary).
Time Frame: Baseline, 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2624803 1 mg | LY2624803 3 mg | Zolpidem 5 or 10 mg | Placebo
Number analyzed (Participants) | 102 | 102 | 102 | 101
units on a scale
  Total Score | 0.17 (0.035) | 0.17 (0.034) | 0.25 (0.034) | 0.13 (0.034)
  Feeling upon Awakening Subscale | 0.14 (0.034) | 0.13 (0.033) | 0.19 (0.033) | 0.12 (0.033)
  Sleep Experience Subscale | 0.22 (0.042) | 0.24 (0.042) | 0.35 (0.042) | 0.15 (0.041)

7. Secondary Outcome: Change From Baseline in Participants' Impression of Daytime Functioning Measured by Daily Consequences of Insomnia Questionnaire (DCIQ) at Week 4 (Week 2 of Period B) Endpoint
Description: DCIQ scale is asked in the participant-reported daily evening questionnaire; 5 point Likert scale with minimum of 0 and maximum of 44 (the higher the score, the more consequences of insomnia). Scale is averaged across study Period B (2 weeks). Change score subtracts Period B average from Period A average (baseline). ANCOVA Model with dependent variable being change from baseline scores and independent variables being treatment, baseline, age group (<65 or ≥65), and insomnia type (primary vs. secondary).
Time Frame: Baseline, 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2624803 1 mg | LY2624803 3 mg | Zolpidem 5 or 10 mg | Placebo
Number analyzed (Participants) | 100 | 99 | 96 | 97
units on a scale | -1.23 (0.395) | -0.87 (0.385) | -1.20 (0.394) | -0.73 (0.386)

8. Secondary Outcome: Change From Baseline in the Insomnia Severity Index (ISI) at Week 4 (Week 2 of Period B) Endpoint
Description: The ISI is a brief self-report instrument that measures a participant's perception of his or her insomnia. 7 questions on 5-point Likert scale with minimum of 0 and maximum of 28. The higher the score, the more severe the insomnia. It was collected at the bi-weekly office visits. ANCOVA Model with dependent variable being change from baseline scores and independent variables being treatment, baseline, age group (<65 or ≥65), and insomnia type (primary vs. secondary).
Time Frame: Baseline, 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2624803 1 mg | LY2624803 3 mg | Zolpidem 5 or 10 mg | Placebo
Number analyzed (Participants) | 99 | 96 | 95 | 94
units on a scale | -2.85 (0.587) | -2.83 (0.578) | -4.63 (0.582) | -1.95 (0.574)

9. Secondary Outcome: Change From Baseline in Physical and Mental Component Scores as Measured by the Short Form 12 (SF-12) Version 2 at Week 4 (Week 2 of Period B) Endpoint
Description: The SF-12 is a subset of 12 items from the Medical Outcomes Study 36-Item Short Form Survey (SF-36) and was collected at the bi-weekly office visits. Each score ranges from 0-100. The components measure physical and mental health, respectively. Higher scores are indicative of better function. ANCOVA Model with dependent variable being change from baseline scores and independent variables being treatment, baseline, age group (<65 or ≥65), and insomnia type (primary vs. secondary)
Time Frame: Baseline, 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2624803 1 mg | LY2624803 3 mg | Zolpidem 5 or 10 mg | Placebo
Number analyzed (Participants) | 97 | 95 | 94 | 92
units on a scale
  Physical Component Scores | -2.32 (1.001) | -0.28 (0.987) | -0.82 (0.992) | -1.84 (0.991)
  Mental Component Scores | 2.49 (1.198) | 1.11 (1.181) | 1.21 (1.191) | 1.94 (1.184)

10. Secondary Outcome: Change From Baseline in Health-related Quality of Life as Measured by European Quality of Life (EuroQol) at Week 4 (Week 2 of Period B) Endpoint
Description: The EuroQoL Questionnaire-5 Dimension (EQ-5D) is a generic, multidimensional, health-related, quality-of-life instrument. The profile allows participants to rate their health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and mood. The score ranges 0-100. The higher score indicates a better health state perceived by the participant. ANCOVA Model with dependent variable being change from baseline scores and independent variables being treatment, baseline, age group (<65 or ≥65), and insomnia type (primary vs. secondary).
Time Frame: Baseline, 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2624803 1 mg | LY2624803 3 mg | Zolpidem 5 or 10 mg | Placebo
Number analyzed (Participants) | 98 | 95 | 94 | 93
units on a scale | -3.06 (1.525) | -2.56 (1.503) | -1.71 (1.510) | 0.23 (1.503)

11. Secondary Outcome: Treatment Satisfaction as Measured by the Participant Drug Preference Question
Description: After study Periods A, and B, participants were asked to rate their experience with the treatment they had just completed. Data are presented as percentage of participants preferring the treatment received in Period A (placebo) or treatment received in Period B.
Time Frame: Baseline (Period A) and 2 weeks (Period B)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | LY2624803 1 mg | LY2624803 3 mg | Zolpidem 5 or 10 mg | Placebo
Number analyzed (Participants) | 99 | 96 | 95 | 94
percentage of participants
  Period A Treatment (placebo) | 23.2 | 22.9 | 12.6 | 35.1
  Period B Treatment | 76.8 | 77.1 | 87.4 | 64.9

12. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I) in Insomnia at Week 4 (Week 2 of Period B) Endpoint
Description: Measures clinician's perception of participant improvement at the time of assessment compared with the start of treatment. Scores range from 1 (very much improved) to 7 (very much worse). Data are presented as percentage of participants in each category.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | LY2624803 1 mg | LY2624803 3 mg | Zolpidem 5 or 10 mg | Placebo
Number analyzed (Participants) | 102 | 102 | 102 | 99
percentage of participants
  1 - Very much improved | 8.8 | 9.8 | 15.7 | 5.1
  2 - Much improved | 20.6 | 23.5 | 34.3 | 18.2
  3 - Minimally improved | 45.1 | 37.3 | 30.4 | 33.3
  4 - No change | 21.6 | 28.4 | 16.7 | 40.4
  5 - Minimally Worse | 2.0 | 0 | 1.0 | 3.0
  6 - Much worse | 2.0 | 1.0 | 2.0 | 0
  7 - Very much worse | 0 | 0 | 0 | 0

13. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) in Insomnia at Week 4 (Week 2 of Period B) Endpoint
Description: A scale that measures the participant's perception of improvement at the time of assessment compared with the start of treatment. The score ranges from 1 (very much improved) to 7 (very much worse). Data are presented as percentage of participants in each category.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | LY2624803 1 mg | LY2624803 3 mg | Zolpidem 5 or 10 mg | Placebo
Number analyzed (Participants) | 99 | 96 | 95 | 94
percentage of participants
  1 - Very much improved | 0 | 2.1 | 4.2 | 3.2
  2 - Much improved | 11.1 | 16.7 | 20.0 | 9.6
  3 - Minimally improved | 62.6 | 45.8 | 55.8 | 42.6
  4 - No change | 24.2 | 31.3 | 15.8 | 37.2
  5 - Minimally worse | 1.0 | 2.1 | 4.2 | 6.4
  6 - Much worse | 0 | 1.0 | 0 | 1.1
  7 - Very much worse | 1.0 | 1.0 | 0 | 0

14. Secondary Outcome: Change From Baseline in Total Sleep Time at Week 4 (Week 2 of Period B) Endpoint Based on Insomnia Type
Description: Total Sleep Time is defined as time in bed minus total time awake. Minimum would be 0; no defined maximum (except if as defined as time in bed). The higher the number, the more time asleep. Analyses were not performed by insomnia type (primary versus secondary) as originally planned because of insufficient number of secondary insomnia participants.
Time Frame: Baseline, 2 weeks
Population: Analyses were not performed by insomnia type because of insufficient number of secondary insomnia patients. Zero participants were analyzed.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | LY2624803 1 mg | LY2624803 3 mg | Zolpidem 5 or 10 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) Based on Insomnia Type
Description: Number of participants with AEs and SAEs. Analyses were not performed by insomnia type (primary versus secondary) as originally planned because of insufficient number of secondary insomnia participants.
Time Frame: Baseline through 8 weeks
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | LY2624803 1 mg | LY2624803 3 mg | Zolpidem 5 or 10 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

16. Secondary Outcome: Change From Baseline in Total Sleep Time at Week 4 (Week 2 of Period B) Endpoint Based on Age Group
Description: Total Sleep Time is defined as time in bed minus total time awake. Minimum would be 0; no defined maximum (except if as defined as time in bed). The higher the number, the more time asleep. Analyses were not performed by age group (under age 65 versus over age 65) as originally planned because of insufficient number of elderly participants.
Time Frame: Baseline, 2 weeks
Population: Analyses were not performed by age group because of insufficient number of elderly patients. Zero participants were analyzed.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | LY2624803 1 mg | LY2624803 3 mg | Zolpidem 5 or 10 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) Based on Age Group
Description: Number of participants with AEs and SAEs. Analyses were not performed by age group (under age 65 versus over age 65) as originally planned because of insufficient number of elderly participants.
Time Frame: Baseline through 8 weeks
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: participants
Arm/Group | LY2624803 1 mg | LY2624803 3 mg | Zolpidem 5 or 10 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

18. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE)
Description: Treatment Emergent Adverse Events (TEAEs) are defined as AEs that first occurred or worsened during the treatment period. TEAEs are summarized by study period and treatment group. TEAEs do not distinguish whether the events were deemed serious. A summary of non-serious AEs is located in the Reported Adverse Event module.
Time Frame: Baseline through 8 weeks
Population: All randomized Cohorts 1 and 2 participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | LY2624803 1 mg | LY2624803 3 mg | Zolpidem 5 or 10 mg | Placebo
Number analyzed (Participants) | 114 | 113 | 117 | 117
participants
  Period B (n= 114, 113, 117, 117) | 28 | 18 | 33 | 21
  Period C (n= 103, 97, 97, 98) | 26 | 34 | 42 | 22
  Period D (n= 91, 89, 94, 88) | 29 | 35 | 34 | 25

19. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: SAEs do not distinguish whether the events are treatment-emergent. A summary of SAEs is located in the Reported Adverse Event module.
Time Frame: Baseline through 8 weeks
Population: All randomized Cohorts 1 and 2 participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | LY2624803 1 mg | LY2624803 3 mg | Zolpidem 5 or 10 mg | Placebo
Number analyzed (Participants) | 114 | 113 | 117 | 117
participants | 1 | 1 | 2 | 2

20. Secondary Outcome: Change From Baseline in Blood Pressure (BP) at Each 2-Week Treatment Endpoint
Description: Change from baseline to the end of each of the 2-week treatment periods (Periods B, C, and D) for systolic blood pressure (SBP) and diastolic blood pressure (DBP) are presented. Least Squares Mean (LSMean) values were adjusted for baseline and treatment.
Time Frame: Baseline, 2 weeks of treatment over 8 weeks
Population: All randomized Cohorts 1 and 2 participants who received at least one dose of study drug, and had both baseline and endpoint values.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LY2624803 1 mg | LY2624803 3 mg | Zolpidem 5 or 10 mg | Placebo
Number analyzed (Participants) | 114 | 113 | 117 | 117
mmHg
  Period B: DBP (n= 112, 111, 117, 117) | 0.15 (0.607) | 0.21 (0.610) | -0.45 (0.594) | -0.41 (0.594)
  Period B: SBP (n= 112, 111, 117, 117) | 0.83 (0.908) | 0.91 (0.912) | -0.05 (0.888) | -0.37 (0.888)
  Period C: DBP (n= 102, 97, 97, 97) | 0.35 (0.675) | 1.11 (0.693) | -0.68 (0.693) | -0.51 (0.693)
  Period C: SBP (n= 102, 97, 97, 97) | 2.31 (0.932) | 1.54 (0.960) | 0.68 (0.957) | 0.58 (0.958)
  Period D: DBP (n= 91, 89, 93, 88) | 0.33 (0.751) | -0.31 (0.760) | 0.37 (0.743) | 0.75 (0.764)
  Period D: SBP (n= 91, 89, 93, 88) | 0.03 (1.097) | 1.17 (1.109) | 0.87 (1.085) | 2.39 (1.118)

21. Secondary Outcome: Change From Baseline in Pulse Rate at Each 2-week Treatment Endpoint
Description: Change from baseline to the end of each of the 2-week treatment periods (Periods B, C, and D) for pulse rate are presented. Least Squares Mean (LSMean) values were adjusted for baseline and treatment.
Time Frame: Baseline, 2 weeks of treatment over 8 weeks
Population: as for outcome 20
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | LY2624803 1 mg | LY2624803 3 mg | Zolpidem 5 or 10 mg | Placebo
Number analyzed (Participants) | 114 | 113 | 117 | 117
beats per minute
  Period B (n= 112, 111, 117, 117) | 0.65 (0.664) | 0.95 (0.669) | 0.41 (0.653) | 0.62 (0.649)
  Period C (n= 102, 97, 97, 97) | 0.42 (0.758) | 0.94 (0.777) | -0.64 (0.777) | -0.02 (0.777)
  Period D (n= 91, 89, 93, 88) | 0.48 (0.813) | -0.36 (0.820) | 1.49 (0.803) | 1.40 (0.826)

22. Secondary Outcome: Change From Baseline in Weight at Each 2-week Treatment Endpoint
Description: Change from baseline to the end of each of the 2-week treatment periods (Periods B, C, and D) for body weight are presented. Least Squares Mean (LSMean) values were adjusted for baseline and treatment.
Time Frame: Baseline, 2 weeks of treatment over 8 weeks
Population: as for outcome 20
Measure: Least Squares Mean (Standard Error); unit: kilogram
Arm/Group | LY2624803 1 mg | LY2624803 3 mg | Zolpidem 5 or 10 mg | Placebo
Number analyzed (Participants) | 114 | 113 | 117 | 117
kilogram
  Period B (n= 111, 111, 115, 114) | 0.13 (0.105) | 0.27 (0.105) | -0.08 (0.103) | 0.06 (0.104)
  Period C (n= 104, 100, 97, 96) | 0.03 (0.129) | 0.30 (0.132) | -0.07 (0.135) | 0.09 (0.134)
  Period D (n=91, 90, 93, 88) | 0.12 (0.164) | 0.17 (0.165) | 0.08 (0.162) | 0.03 (0.166)

23. Secondary Outcome: Number of Participants With Abnormal Laboratory Analytes at Each 2-Week Treatment Endpoint
Description: Summary of number of participants with abnormal clinical chemistry, hematology and urinalysis laboratory results. A participant is included in the abnormal category if he/she experienced a result outside the normal reference ranges based on Lilly's reference range in the current period. All analytes have both lower and upper limits. The abnormal number includes both low (below normal range) and high (above normal range).
Time Frame: 2 weeks of treatment over 8 weeks
Population: All randomized Cohorts 1 and 2 participants who received at least one dose of study drug, and had endpoint value. For LY2624803 1 mg, LY2624803 3 mg, Zolpidem 5 or 10 mg, and Placebo, the Number of Participants Analyzed were as follows: Period B: N=114, 113,117, 117; Period C: N=103, 97, 97, 98; and Period D: N=91, 89, 94, 88.
Measure: Number; unit: participants
Arm/Group | LY2624803 1 mg | LY2624803 3 mg | Zolpidem 5 or 10 mg | Placebo
Number analyzed (Participants) | 114 | 113 | 117 | 117
participants
  Period B: Alkaline Phosphatase | 0 | 1 | 0 | 0
  Period B: Alanine Transaminase | 1 | 0 | 1 | 0
  Period B: Aspartate Transaminase | 1 | 1 | 0 | 0
  Period B: Total Bilirubin | 1 | 2 | 0 | 2
  Period B: Creatine Phosphokinase | 1 | 3 | 2 | 4
  Period B: Creatinine | 3 | 1 | 4 | 5
  Period B: Glucose, Non-fasting or random | 6 | 4 | 2 | 3
  Period B: Blood Urea Nitrogen | 2 | 1 | 2 | 2
  Period B: Hemoglobin | 2 | 1 | 0 | 1
  Period B: Leukocyte Count | 2 | 1 | 2 | 0
  Period B: Platelet Count | 1 | 1 | 1 | 0
  Period C: Alkaline Phosphatase | 0 | 0 | 0 | 0
  Period C: Alanine Transaminase | 0 | 0 | 2 | 1
  Period C: Aspartate Transaminase | 0 | 0 | 0 | 0
  Period C: Total Bilirubin | 1 | 1 | 2 | 1
  Period C: Creatine Phosphokinase | 3 | 2 | 0 | 2
  Period C: Creatinine | 3 | 0 | 4 | 3
  Period C: Glucose, Non-fasting or random | 4 | 5 | 1 | 5
  Period C: Blood Urea Nitrogen | 2 | 2 | 1 | 3
  Period C: Hemoglobin | 1 | 0 | 2 | 0
  Period C: Leukocyte Count | 2 | 3 | 0 | 1
  Period C: Platelet Count | 1 | 0 | 1 | 0
  Period D: Alkaline Phosphatase | 0 | 0 | 0 | 0
  Period D: Alanine Transaminase | 0 | 1 | 1 | 0
  Period D: Aspartate Transaminase | 2 | 1 | 1 | 1
  Period D: Total Bilirubin | 3 | 1 | 1 | 0
  Period D: Creatine Phosphokinase | 2 | 2 | 5 | 1
  Period D: Creatinine | 1 | 4 | 4 | 2
  Period D: Glucose, Non-fasting or random | 6 | 2 | 4 | 2
  Period D: Blood Urea Nitrogen | 0 | 2 | 0 | 1
  Period D: Hemoglobin | 0 | 1 | 0 | 2
  Period D: Leukocyte Count | 1 | 2 | 3 | 5
  Period D: Platelet Count | 0 | 3 | 0 | 1

24. Secondary Outcome: Change From Baseline in Heart Rate as Measured by Electrocardiogram (ECG) at Each 2-week Treatment Endpoint
Description: Change from baseline to the end of each of the 2-week treatment periods (Periods B, C, and D) for heart rate are presented. Least Squares Mean (LSMean) values were adjusted for baseline and treatment.
Time Frame: Baseline, 2 weeks of treatment over 8 weeks
Population: All randomized Cohort 1 and 2 participants who received at least one dose of study drug, and had both baseline and endpoint values.
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | LY2624803 1 mg | LY2624803 3 mg | Zolpidem 5 or 10 mg | Placebo
Number analyzed (Participants) | 114 | 113 | 117 | 117
beats per minute
  Period B (n= 112, 110, 115, 112) | 1.09 (0.689) | 0.26 (0.695) | 1.10 (0.681) | 0.30 (0.688)
  Period C (n= 99, 94, 96, 95) | -0.59 (0.734) | 0.31 (0.753) | -0.02 (0.745) | 1.14 (0.749)
  Period D (n= 91,86, 93, 87) | 1.71 (0.827) | 1.71 (0.851) | 1.43 (0.818) | 0.86 (0.846)

25. Secondary Outcome: Change From Baseline in QT Interval Corrected Using Fridericia Formula (QTcF) as Measured by Electrocardiogram (ECG) at Each 2-week Treatment Endpoint
Description: QT interval is a measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle. QTcF is the QT interval corrected for heart rate using Fridericia formula. Least Squares Mean (LSMean) values were adjusted for baseline and treatment.
Time Frame: Baseline, 2 weeks of treatment over 8 weeks
Population: as for outcome 24
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Arm/Group | LY2624803 1 mg | LY2624803 3 mg | Zolpidem 5 or 10 mg | Placebo
Number analyzed (Participants) | 114 | 113 | 117 | 117
milliseconds
  Period B (n= 112, 110, 115, 112) | -0.04 (1.314) | -2.62 (1.325) | -1.02 (1.300) | -1.43 (1.316)
  Period C (n= 99, 94, 96, 95) | -1.07 (1.335) | -0.41 (1.373) | -3.27 (1.356) | -3.92 (1.370)
  Period D (n= 91, 86, 93, 87) | -2.00 (1.319) | -2.99 (1.344) | -3.59 (1.293) | -1.68 (1.339)

ADVERSE EVENTS:
Time Frame: Adverse events are reported for periods B, C, and D. The number of participants at risk vary depending upon the period in which the AE occurred. Due to discontinuations, later periods had fewer participants.
Groups:
- Period B - LY2624803 1 mg: Patients received LY2624803 1 mg in Period B (2-week treatment period.
- Period B - LY2624803 3 mg: Patients received LY2624803 3 mg in Period B (2-week treatment period).
- Period B - Placebo: Patients received placebo in Period B (2-week treatment period).
- Period B - Zolpidem 5 or 10 mg: Patients received Zolpidem 5 or 10 mg in Period B (2-week treatment period).
- Period C - LY2624803 1 mg: Patients received LY2624803 1 mg in Period C (2-week treatment period.
- Period C - LY2624803 3 mg: Patients received LY2624803 3 mg in Period C (2-week treatment period).
- Period C - Placebo: Patients received placebo in Period C (2-week treatment period).
- Period C - Zolpidem 5 or 10 mg: Patients received Zolpidem 5 or 10 mg in Period C (2-week treatment period).
- Period D - LY2624803 1 mg: Patients received LY2624803 1 mg in Period D (2-week treatment period.
- Period D - LY2624803 3 mg: Patients received LY2624803 3 mg in Period D (2-week treatment period).
- Period D - Placebo: Patients received placebo in Period D (2-week treatment period).
- Period D - Zolpidem 5 or 10 mg: Patients received Zolpidem 5 or 10 mg in Period D (2-week treatment period).
Arm/Group | Period B - LY2624803 1 mg | Period B - LY2624803 3 mg | Period B - Placebo | Period B - Zolpidem 5 or 10 mg | Period C - LY2624803 1 mg | Period C - LY2624803 3 mg | Period C - Placebo | Period C - Zolpidem 5 or 10 mg | Period D - LY2624803 1 mg | Period D - LY2624803 3 mg | Period D - Placebo | Period D - Zolpidem 5 or 10 mg
Serious Adverse Events (participants affected / at risk) | 1/114 | 1/113 | 0/117 | 1/117 | 0/103 | 0/97 | 2/98 | 1/97 | 0/91 | 0/89 | 0/88 | 0/94
Other Adverse Events (participants affected / at risk) | 28/114 | 18/113 | 21/117 | 33/117 | 26/103 | 34/97 | 22/98 | 42/97 | 29/91 | 35/89 | 25/88 | 34/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period B - LY2624803 1 mg (N=114) | Period B - LY2624803 3 mg (N=113) | Period B - Placebo (N=117) | Period B - Zolpidem 5 or 10 mg (N=117) | Period C - LY2624803 1 mg (N=103) | Period C - LY2624803 3 mg (N=97) | Period C - Placebo (N=98) | Period C - Zolpidem 5 or 10 mg (N=97) | Period D - LY2624803 1 mg (N=91) | Period D - LY2624803 3 mg (N=89) | Period D - Placebo (N=88) | Period D - Zolpidem 5 or 10 mg (N=94)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period B - LY2624803 1 mg (N=114) | Period B - LY2624803 3 mg (N=113) | Period B - Placebo (N=117) | Period B - Zolpidem 5 or 10 mg (N=117) | Period C - LY2624803 1 mg (N=103) | Period C - LY2624803 3 mg (N=97) | Period C - Placebo (N=98) | Period C - Zolpidem 5 or 10 mg (N=97) | Period D - LY2624803 1 mg (N=91) | Period D - LY2624803 3 mg (N=89) | Period D - Placebo (N=88) | Period D - Zolpidem 5 or 10 mg (N=94)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Stomach discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Feeling abnormal (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling jittery (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sluggishness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suprapubic pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 4 (4) | 3 (3) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram t wave abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coordination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Dizziness exertional (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (6) | 1 (1) | 3 (3) | 2 (3) | 3 (3) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 2 (2) | 2 (2) | 6 (6)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sedation (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Sleep paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 5 (5) | 4 (4) | 6 (6) | 3 (3) | 7 (7) | 7 (7) | 2 (2) | 3 (3) | 4 (4)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypervigilance (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Initial insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep inertia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine spasm (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postmenopause (Social circumstances) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days